CLINICAL TRIAL: NCT00609453
Title: Brain Imaging of Psychotherapy for Depression (Includes, "Reward System Recovery Following Behavioral Activation Therapy in Depression")
Brief Title: Brain Imaging of Psychotherapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Gabriel Dichter, Associate Professor of Psychiatry, University of North Carolina, Chapel Hill
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 05-2605; NIMH R03 MH078145
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Major Depressive Disorder
Keywords: Control participants
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Individuals with major depressive disorder receiving therapy
  Interventions: Behavioral: Brief Behavioral Activation Treatment for Depression

INTERVENTIONS:
Behavioral: Brief Behavioral Activation Treatment for Depression — Weekly individual therapy sessions

SUMMARY:
The goal of the proposed research is to examine the neural correlates of depressive symptom reduction in individuals with major depressive disorder using functional magnetic resonance imaging (fMRI), and to compare results to those obtained from a nondepressed control group.

ELIGIBILITY:
Inclusion Criteria:

* For group 1: Diagnosis of current depression and no other current Axis I psychiatric disorder
* For group 1: Hamilton Depression Rating Scale score of 15 or greater

Exclusion Criteria:

* A history of serious head injury or neurological disease or psychosis
* Current use of psychoactive medications
* Factors that could affect MRI safety including current or planned pregnancy
* For group 2: current Axis I psychiatric disorder, as assessed by structured clinical interview

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Inventory | three times over 12 weeks
Functional Magnetic Resonance Imaging | twice in 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel S Dichter, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Duke-UNC Brain Imaging and Analysis Center, Durham, North Carolina, United States